CLINICAL TRIAL: NCT06361693
Title: "Observational Descriptive Study of Patient-performed Preoxygenation, the "Autopreoxygenation Concept""
Brief Title: Descriptive Observational Study of Patient-performed Pre-oxygenation
Acronym: ApréOx
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240147; 2024-A00143-44 (Other: France : Ministry of Health)
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-09

CONDITIONS: Anesthesia; ASA Physical Status I; ASA Physical Status II
Keywords: Preoxygenation; General anesthesia; Adult; Preoperative anxiety
MeSH Terms: interventions — argipressin, Asu(1,6)-

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Adult patients benefiting from planned outpatient surgery under general anesthesia.
  Interventions: Other: Auto-preoxygenation; Other: APAIS scale; Other: Visual analog anxiety scale (VAS-A); Other: Visual analog comfort scale (VAS-C)

INTERVENTIONS:
Other: Auto-preoxygenation — Management is not modified. Routine monitoring (ECG, BP, SpO2). As in care, the patient takes the mask and the respirator is started, delivering an inspired oxygen fraction of 100% (FiO2=1).
  Monitoring of : inspired fraction of oxygen, expired fraction of oxygen and end-tidal fraction of carbon dioxide. The ventilator also provides the respiratory rate and tidal volume carried out by the patient.
  The fresh gas flow is set by default and will be adjusted to 12l/min for patient comfort.After less than a minute, a normal capnia curve and the presence of an FeO2 value appear. Here, time is standardized to 1 min. In the absence of one of these elements, the caregiver always takes control of preoxygenation.Timer is started, it is T0 min. At T 3min, collection of values and decision-making :
  * objectives achieved : end of this sequence.
  * objectives not achieved, the caregiver takes control again for an additional 2 minutes in order to seek to achieve an FeO2>90%.
Other: APAIS scale — APAIS scale
Other: Visual analog anxiety scale (VAS-A) — Visual analog anxiety scale (VAS-A)
Other: Visual analog comfort scale (VAS-C) — Visual analog comfort scale (VAS-C)

SUMMARY:
The aim of this research would be to determine the efficacy and effects of preoxygenation when performed by the patient (mask held by the patient).

This is the concept of "self-preoxygenation".

DETAILED DESCRIPTION:
Pre-oxygenation is a fundamental element of the induction sequence in anesthesia, described and recommended since 1955. Numerous studies have examined and compared the various techniques for implementing this procedure in terms of duration, objectives, equipment, patient characteristics and conditions. None of them specifies who should hold the mask when carrying out this recommendation. In everyday practice, patients are often asked to hold the mask themselves. A preliminary survey showed that 86% of patients are offered this option. The professionals questioned cited relational reasons (83%) above all, but also organizational reasons (43%).

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing scheduled surgery with general anesthesia
* Patient classified ASA I or II
* Patient understanding and speaking French
* Patient informed of the study and not opposed to it
* Decision to have preoxygenation carried out by the patient.

Exclusion Criteria:

* Patients with grade II or III obesity (BMI>35)
* Patient with at least one respiratory comorbidity
* Smoking patient
* Pregnant patients
* Patient with an allergy to one of the mask's components
* Patient with cognitive impairment or known comprehension difficulties
* Patient under guardianship or curatorship
* Patient not affiliated to health care system

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major patient (adults) undergoing scheduled outpatient surgery requiring general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
FeO2>90% | 3 minuts after the beginning of auto-preoxygenation - Day 1
  Percentage of patients achieving a FeO2>90% in 3 min at 12L/min fresh gas flow on 100% oxygen.
  To Evaluate the efficacity of the self-preoxygenation Assessing the effectiveness of auto-preoxygenation

SECONDARY OUTCOMES:
APAIS anxiety score | At arrival in the Day Surgery Unit - Day 1
  Percentage of patients with a total APAIS anxiety score greater than 10/20 in women, 12/20 in men on arrival in the operating room
Visual analog anxiety scale (VAS-A) score | At arrival in the Day Surgery Unit - Day 1
  Percentage of patients with a decrease in the visual analog anxiety scale score (VAS-A) between arrival and discharge in the Day Surgery Unit.
  Assessing the effect of self-preoxygenation on preoperative anxiety
Visual analog anxiety scale (VAS-A) score | At discharge from the Day Surgery Unit - Day 1
  Percentage of patients with a decrease in the visual analog anxiety scale score (VAS-A) between arrival and discharge in the Day Surgery Unit.
  Assessing the effect of self-preoxygenation on preoperative anxiety
Visual analog comfort scale (VAS-C) score | At discharge from the Day Surgery Unit - Day 1
  Percentage of patients having obtained a visual analog comfort scale (VAS-C) score greater than 5 out of 10 upon discharge from the Day Surgery Unit.
  Assessing the effect of self-preoxygenation on comfort

CONTACTS AND LOCATIONS:
Overall Officials: Sophie TOUSSAINT, Nurse anesthetist, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Anesthesia-intensive care department - Cochin - Port-Royal hospital - APHP, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No